CLINICAL TRIAL: NCT06348420
Title: Anti-reflux Mucosal Valvuloplasty Versus Proton Pump Inhibitors for the Treatment of Patients With Gastroesophageal Reflux Disease in a Tertiary Healthcare Center in China: Study Protocol for a Randomized Controlled Trial
Brief Title: Anti-reflux Mucosal Valvuloplasty Versus PPIs for GERD Treatment
Acronym: ARMV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Lu Jiaoyang, professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-QILU-LU 03
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Endoscopic anti-reflux; Proton pump inhibitor; Randomized controlled trial; Gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARMV (intervention group) (Experimental): Under general anesthesia, patients are positioned in the left lateral decubitus position and undergo endoscopic examination of the esophagus and stomach. The surgery utilizes a single-channel gastroscope (EG29-i10, Pentax, Japan, or GIF-H290T, Olympus, Japan) and a high-frequency generator (VIO300D, Erbe, Germany). A transparent cap (D-201, Olympus, Japan) is attached to the gastroscope to improve visualization and aid in manipulating the flap valve. The DualKnife (Olympus, Japan) is selected for dissection due to its maneuverability in a retroflexed fashion. For patients with esophageal strictures obstructing scope passage, esophageal dilation is performed using Savary-Gilliard dilators (Cook Medical, USA) just before ARMV.
  Interventions: Procedure: anti-reflux mucosal valvuloplasty (ARMV)
- PPI (control group) (No Intervention): Patients randomized to the PPI group will follow the PPI treatment scheme. If GERD symptoms are effectively controlled with their current PPI dosage for at least one month, the regimen is decreased by one step. Conversely, if symptoms are poorly controlled, the dosage is increased by one step based on the PPI algorithm, which aligns with best clinical practices. The use of PPI will be recorded in medication diaries using generic names listed in the table below and classified according to the daily dose and frequency. Dosage will be categorized as "double dose" = ≥30 or 40 mg per day, "full dose" = 30 or 40 mg per day, "half dose" = 15 or 20 mg per day, "occasional" or "on demand" = < "full dose" taken for < 50% of days in the follow-up period. Common medications include Nexium 20mg、Prevacid 30mg、Prilosec 20mg、Protonix 20mg、Aciphex20mg.The frequency of medication use is once a day.

INTERVENTIONS:
Procedure: anti-reflux mucosal valvuloplasty (ARMV) — During the ARMV procedure, a segment of the mucosa at the esophagogastric junction (EGJ) is released and reconstructed to form a mucosal flap. Cautery markings are made on 3/4-4/5 of the mucosa along the lesser curvature, approximately 2 cm below the dentate line. After submucosal injection of saline with indigocarmine, the premarked mucosa is dissected from the caudal to cranial side using an endoscopic submucosal dissection technique. The cranial edge of the released mucosa is left in place, and the semi-free mucosa naturally curls to form a double-layer flap. Metal clips are then used to anchor the free edge of the mucosa to the exposed submucosa/smooth muscle to prevent flattening of the mucosal flap. Any visible bleeding on the exposed submucosa is coagulated using electric forceps.
  Arms: ARMV (intervention group)

SUMMARY:
The study objective is to evaluate the relative merits, safety and effectiveness of Anti-reflux mucosal valvuloplasty (ARMV) in GERD patients currently treated with daily Proton Pump Inhibitors (PPIs).

DETAILED DESCRIPTION:
Under general anesthesia, patients are positioned in the left lateral decubitus position and undergo endoscopic examination of the esophagus and stomach. The surgery utilizes a single-channel gastroscope (EG29-i10, Pentax, Japan, or GIF-H290T, Olympus, Japan) and a high-frequency generator (VIO300D, Erbe, Germany). A transparent cap (D-201, Olympus, Japan) is attached to the gastroscope to improve visualization and aid in manipulating the flap valve. The DualKnife (Olympus, Japan) is selected for dissection due to its maneuverability in a retroflexed fashion. For patients with esophageal strictures obstructing scope passage, esophageal dilation is performed using Savary-Gilliard dilators (Cook Medical, USA) just before ARMV.

During the ARMV procedure, a segment of the mucosa at the esophagogastric junction (EGJ) is released and reconstructed to form a mucosal flap. Cautery markings are made on 3/4-4/5 of the mucosa along the lesser curvature, approximately 2 cm below the dentate line. After submucosal injection of saline with indigocarmine, the premarked mucosa is dissected from the caudal to cranial side using an endoscopic submucosal dissection technique. The cranial edge of the released mucosa is left in place, and the semi-free mucosa naturally curls to form a double-layer flap. Metal clips are then used to anchor the free edge of the mucosa to the exposed submucosa/smooth muscle to prevent flattening of the mucosal flap. Any visible bleeding on the exposed submucosa is coagulated using electric forceps.

After the ARMV procedure, PPI therapy is continued for 1 month to promote mucosal healing before being discontinued. If symptoms reoccur, the PPI management regimen is reinstated for the ARMV group, with diligent recording of PPI usage in a medication diary.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age;
* Hiatal hernia ≤ 2 cm;
* Sliding hernia ≤ 2 cm;
* Recurrence of GERD symptoms after cessation of PPIs;
* On daily PPI for ≥1 year or twice daily PPI for at least 8 weeks;
* Esophagitis (Los Angeles Classification) Grade B, C, or D;
* Hill's flap valve grade ≤ III;
* Observation of distal esophageal pH < 4 on at least 1-2 days within a 7-day period, with a percentage exceeding 5.3%;
* Normal or near-normal esophageal motility;
* Lower esophageal sphincter pressure (LESP) ranging between 5-15 mmHg;
* DeMeester score ≥ 14.7 or total reflux episodes exceeding 73;
* Completion of a signed informed consent form.

Exclusion Criteria:

* BMI > 35 kg/m2;
* ASA > II;
* Barrett's esophagus;
* Hiatal hernia > 2 cm;
* Esophagitis (Los Angeles Classification) Grade A or No esophagitis；
* Hill's flap valve grade > III；
* Peptic ulcer disease;
* Primary esophageal motility disorders such as achalasia;
* Severe gastroparesis;
* History of previous esophageal or gastric surgery, including ARMS or ARMA;
* Uncontrolled systemic diseases;
* Gastric outlet obstruction;
* Pregnancy or planning to become pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
GERD-HRQL | at 0, 6 months follow- up
  Questionnaire (GERD-HRQL) : Total Score: Calculated by summing the individual scores to questions 1-15 Greatest possible score (worst symptoms)= 75 Lowest possible score (no symptoms)= 0 Heartburn Score: Calculated by summing the individual scores to questions 1-6 . Worst heartburn symptoms = 30 No heartburn symptoms= 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination. Regurgitation Score: Calculated by summing the individual scores to questions10-15. Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

SECONDARY OUTCOMES:
GERD-Q score | at 0, 3, 6 ,12 ,24,36 months follow- up
  Questionnaire (GERD-Q ) : Recall the frequency of burning sensation (heartburn) after your sternum in the past 7 days;How often do you feel stomach contents (liquid or food) returning to your throat or mouth (reflux) in the past 7 days?How often did you feel pain in the center of your upper abdomen in the past 7 days?How often did you feel nauseous in the past 7 days?How often have you had difficulty getting good night sleep due to heartburn and/or reflux in the past 7 days? Looking back on the past 7 days, in addition to the medication advised by the doctor, did you take additional medication to alleviate the frequency of heartburn and/or reflux? (such as calcium carbonate, aluminum hydroxide, and other antacids).0 days are 0 points, 1 day is 1 point, 2-3 days are 2 points, and 4-7 days are 3 points. Add up the scores for each item to obtain the total score.
DeMeester score | at 0, 6 and 24 months follow- up
  Esophageal 24-hintraluminal ambulatory pH monitoring is performed to monitor the modality of the reflux. A catheter sensor is placed 5 cm above the proximal border of the lower esophageal sphincter (LES). Each reflux is considered acidic when the pH of the refluxate is less than 4. The acid reflux composite score (DeMeester score) is calculated using the following values: percentage of total time in reflux, percentage of time in reflux in the upright position, percentage of time in reflux in the supine position, the total number of reflux episodes, number of reflux episodes continuing over 5 minutes, and longest duration of reflux among all reflux episodes
Presence of reflux esophagitis | at 0, 6 and 24 months follow- up
  Healing of esophagitis will represent a clinically significant improvement. Treatment success will be defined by a significantly (p < 0.05) higher number of patients with healed esophagitis in the ARMV group vs. PPI group.
Appearance of the mucosal flap | at 6 and 24 months follow- up
  The shape and mobility of the anti-reflux mucosal flap displayed under endoscopy
PPI use | at 0, 3, 6 ,12 ,24,36 months follow- up
  Requirement of PPI for control of symptoms. Heartburn and Regurgitation questionnaire 0 =No symptom 1 =Symptoms noticeable but not bothersome 2=Symptoms noticeable and bothersome but not every day 3 =Symptoms bothersome every day 4 =Symptoms affect daily activity 5 =Symptoms are incapacitating to do daily activities.
Incidence of adverse events | at 3, 6 ,12 ,24,36 months follow- up
  The incidence of intraoperative and postoperative bleeding and perforation; Postoperative pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Department of Gastroenterology and Endoscopy Center, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
We do not currently plan to grant public access to the participant-level dataset due to privacy concerns and data protection regulations. However, data access may be considered upon reasonable request, subject to ethical and regulatory approvals, to ensure compliance with participant confidentiality and legal requirements.

REFERENCES:
- [Derived] Lv X, Ma W, Zeng Y, Lu J. Antireflux mucosal valvuloplasty versus proton pump inhibitors for the treatment of patients with gastro-oesophageal reflux disease in a tertiary healthcare centre in China: study protocol for a randomised controlled trial. BMJ Open. 2024 Dec 22;14(12):e088970. doi: 10.1136/bmjopen-2024-088970. PMID 39773838